CLINICAL TRIAL: NCT03776838
Title: Impact of Nociceptive-Level (NOL) Intraoperative Guided Analgesia on Pain Scores, Opioid Consumption and Recovery in Postoperative Care Unit in Patients Undergoing Gynecological Laparoscopic Surgery Under General Anesthesia. The NOLGYN Pilot Study
Brief Title: Impact of Nociceptive-Level (NOL) Intraoperative Guided Analgesia During Gynecological Laparoscopic Surgery Under General Anesthesia
Acronym: NOLGYN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Medasense Biometrics Ltd (Other)
Responsible Party: Principal Investigator, Philippe Richebe, MD PhD, Director of Research, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-1534
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Gynecologic Laparoscopic Surgery; Hysterectomy; Oophorectomy
Keywords: NOL monitoring; anesthesia; fentanyl consumption; intraoperative

STUDY DESIGN:
Intervention Model Description: 2 groups of patients. Randomization into group SoC + NOL vs SoC according to randomization list for a total number of 70 patients
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization into group SoC + NOL vs SoC will be done prior to the entrance in the OR, the day of the surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoC+NOL analgesia guided fentanyl administration (Experimental): A bolus of 2 mcg/kg of IV Fentanyl will be given at the induction of the anesthesia. A bolus of 1 mcg/kg of IV Fentanyl will be given at the time of incision. During surgery, administration of 0.5 mcg/kg of IV Fentanyl will be administered following a pre determinate algorithm based on NOL index + heart rate + mean arterial blood pressure variations.
  Intervention is NOL monitoring in this group that will help to guide intravenous administration of fentanyl during surgery.
  Interventions: Drug: Intravenous Fentanyl guided by SoC+NOL
- SoC analgesia guided group (Active Comparator): A bolus of IV Fentanyl at the discretion of a physician will be given at the induction of the anesthesia. A bolus of IV Fentanyl at the discretion of a physician will be given at the time of incision. During surgery, administration of IV Fentanyl at the discretion of a physician will be administred following a pre determinated algorithm based on heart rate + mean arterial blood pressure variations.
  Intervention will be here to use Heart rate and blood pressure to administer intraoperative intravenous fentanyl.
  Interventions: Drug: Intravenous Fentanyl guided by SoC

INTERVENTIONS:
Drug: Intravenous Fentanyl guided by SoC+NOL — Predeterminated bolus of IV Fentanyl will be given at the induction of anesthesia (2 mcg/kg), at the time of incision (1 mcg/kg). During surgery, administration of 0.5 mcg/kg of IV Fentanyl will be administred following a pre determinated algorithm based on NOL index + heart rate + mean arterial blood pressure variations.
  Arms: SoC+NOL analgesia guided fentanyl administration
Drug: Intravenous Fentanyl guided by SoC — Bolus of IV Fentanyl at the discretion of a physician will be given at the induction of anesthesia, and at the time of incision. During surgery, administration of IV Fentanyl at the discretion of a physician will be administred following a pre determinated algorithm based on heart rate + mean arterial blood pressure variations.
  Arms: SoC analgesia guided group

SUMMARY:
The aim of the present study is to show that the use of the NOL device in addition to the Standard of Care (based on mean arterial blood pressure and heart rate values) to guide the administration of opioids compared to the Standard of Care reduces the total fentanyl consumption and the number of intraoperative administration of IV fentanyl during gynecological laparoscopic surgery and improves postoperative outcomes in PACU.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that the group who will be administered intraoperative fentanyl based on NOL + mean arterial blood pressure (MABP) + heart rate (HR) values (SoC+NOL group) versus on MABP and HR (SoC group) will need less intra and postoperative opioid and will report less postoperative pain which will be reflected by a reduced number of adverse effects associated with opioid and/or reduced postoperative pain scores at the PACU arrival resulting in a faster time of readiness to discharge.

Background: The NOL index, a nociception monitor using a multiparametric approach, has shown an excellent sensitivity and specificity in detecting noxious stimuli under general anesthesia. This monitor is better than any other classically used clinical parameter in grading nociception under general anesthesia. More recently, a strong correlation between NOL index response to nociceptive stimulus and the level of opioid analgesia during surgery was reported. Studies are now conducted in our center (Maisonneuve-Rosemont Hospital, University of Montreal, Montreal, QC, Canada) to show a better post-operative outcome when using intraoperative NOL monitoring to adapt nociception/anti-nociception balance during general anesthesia (GA) for colorectal surgery.

So far, no study has evaluated in gynecological laparoscopic surgery the impact of NOL monitoring to guide the administration of intraoperative IV fentanyl on intra and postoperative opioid consumption and pain scores.

Objectives: Primary objective:

Reduction in total intraoperative fentanyl consumption (in mcg) and number of intraoperative administrations of IV fentanyl in the SoC+NOL analgesia guided versus SoC analgesia guided group (SoC = Standard of Care).

Secondary objectives:

Secondary outcome [1] Post-operative opioid consumption (IV hydromorphone in PACU) until patient is ready for discharge from Post-Anesthesia Care Unit.

Secondary outcome [2] Post-operative pain scores at rest and at coughing recorded in PACU by using numerical pain rating scales (NRS) in PACU (evaluated Q15min for 1h).

Secondary outcome [3] Intraoperative total consumption and frequency of administration of vasoactive drugs.

Secondary outcome [4] Post-operative sedation scores with Ramsay Sedation Score recorded every 15 minutes in PACU for at least 1h Secondary outcome [5]

Post-operative side-effects within 24 hours post-operatively:

1. Nausea and vomiting: measure of the incidence of any nausea, emetic episodes (retching or vomiting), or both (i.e. postoperative nausea and vomiting) during the first 24 postoperative hours. Upon Discharge from PACU, and at 24 hours post-surgery, patients will verbally rate their worst nausea episode since emergence on an 11-point scale, where 0 represented no nausea and 10 the most severe nausea.
2. Respiratory depression: defined as respiratory rate (RR) below 9 respirations per minutes (RPM). Respiratory rate will be recorded at 5-minute intervals, manually or per PACU monitor. The incidence of RR < 9 RPM during the first 1.5 hours since admission to PACU will be recorded, as well as requirement for naloxone reversal of opioids or additional reversal of muscle relaxants.
3. Itching: score of itching recorded every 10-15 minutes on an 11-point scale, where 0 is no itching and 11 is the most severe itching possible.

Secondary outcome [6] Post-operative time to discharge from PACU.

This time will be recorded since it may be different from the actual time of discharge which may be prolonged due to non-medical reasons. Patient discharge will be based upon a or b whichever comes first:

1. Time of readiness to discharge from PACU, based on the evaluation of the Aldrete score (out of 9 points) and patient pain level (HMR local score, out of 16 points).
2. Time of discharge from PACU. Secondary outcome [7] Time to first postoperative pain rescue medication administration in PACU or on wards.

Methods: Enrollment of 70 randomized adult patients undergoing general anesthesia for gynecological laparoscopic surgery (e.g. hysterectomy, uni- or bilateral Oophorectomy), which will be randomized to 2 groups: SoC guided analgesia (control group) versus SoC+NoL guided analgesia (intervention group).

All patients will be consented prior to the surgery. Anesthesia will be standardized for all patients, with: IV lidocaine (0.5mg.kg-1), Propofol (2mg.kg-1), IV fentanyl (2mcg.kg-1), IV rocuronium (0.6mg.kg-1). Depth of anesthesia with sevoflurane will be maintained and monitored with the BIS index kept between 40 and 60. In both the groups, rocuronium will be administered to keep the response to the train of four below 2/4 (TOFScan, Draeger). IV fentanyl will be intraoperatively administered based on HR and MABP variations on the SOC group and HR + MABP + NOL index in the NOL group (see attached decision algorithm). At the end of surgery, all patients will be extubated in the OR, then transferred to PACU. In PACU pain scores and recovery scores (PONV, sedation, respiratory depression, itching, delirium…) and hydromorphone requirements to reach a pain < 3/10 will be assessed as well as Aldrete score and time for readiness for PACU discharge. The study will end at PACU discharge. This study will be registered on clinicaltrial.gov website.

Power calculation: Statistical analyses will be done using SAS version 9.4 or higher and will be performed at a two-sided 0.05 significance level. The primary objective of the study is reduced in total intraoperative fentanyl consumption (in mcg) and number of intraoperative administration of IV fentanyl in the SoC+NOL analgesia guided versus SoC analgesia guided group. Preliminary results from our center (HMR/CEMTL) showed that patients in SOC group had an IV intraoperative fentanyl consumption of 616 +/- 190 mcg during anesthesia. For an expected decrease of 25% in the SoC+NOL group for this PACU IV hydromorphone consumption, with a type I error α = 0.05 (two-tailed), an 90% power, the total sample size needed is 64. To account for an approximative 10% rate of loss to follow-up or missing data due to technical problems, a total of 70 subjects will be recruited. Because of the large number of secondary objectives and to protect against type I error in a less conservative way than the Bonferroni correction, the Holm step-down procedure will be applied to the sets of secondary hypotheses.

Significance/Importance: The main outcomes of this study will be to demonstrate that intraoperative NOL guidance decreases the need of intra- and post-operative opioids and might improve postoperative recovery after this type of gynecological surgery.

Study Design: This is a single-center, prospective, randomized, parallel-group, single-blinded.

Subject Population: Adult patients scheduled to undergo elective gynecological laparoscopic surgery (hysterectomy and uni- or bilateral oophorectomy) under general anesthesia.

Sample Size: 70 patients will be included in this study.

Study Duration: 12 months.

Study Center: Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal (CEMTL), University of Montreal, Montreal, Quebec, Canada.

Adverse Events: None expected.

Subvention: An Independent Investigator Initiated Trial (IIIT) grant application will be sent to the company Medasense Biometrics LTD for the sponsoring of this study. A contract will be made and signed by both the parties: Medasense Biometrics LTD on one hand and the CR-HMR and the CEO of the CEMTL/HMR prior to starting the study.

ELIGIBILITY:
Inclusion Criteria:

1. Female age 18-75 years
2. ASA I-III
3. adult patients scheduled to undergo elective gynecological laparoscopic surgery (hysterectomy and uni- or bilateral oophorectomy) under general anesthesia
4. patient able to consent in the language of the including center

Exclusion Criteria:

1. use of any type of anesthesia other than general anesthesia (neuraxial, epidural analgesia or local regional anesthesia, e.g. transversus abdominal plane block...)
2. patients with non-regular sinus cardiac rhythm, implanted pacemakers, prescirbed antimuscarinic agents, alpha2-adrenergic agonists, beta1-adrenergic antagonists, and antiarrhythmic agents
3. emergent surgery
4. pregnancy/lactation. Pregnancy test will be performed in all women of child bearing age
5. BMI > 35 kg/m2
6. preoperative hemodynamic disturbance
7. central nervous system disorder (neurologic/ head trauma/ uncontrolled epileptic seizures)
8. drug or alcohol abuse within the last 6 months (for women, > 3 drinks on one occasion or >7 drinks during a week)
9. pre-operative chronic opioid use or chronic pain, equivalent to oxycodone 20mg per oral, per day for more than 6 weeks
10. chronic use of psychoactive drugs within 90 days prior to surgery
11. medical conditions qualifying for ASA III or IV:

    1. untreated or persistent peripheral or central cardiovascular disease
    2. severe pulmonary disease e.g. COPD gold 4, FEV< 1.0l/s, or (evidence of) elevated paCO2 > 6.0 kPa
    3. significant hepatic disease with increased bilirubin, INR or low albumin
    4. history of severe cardiac arrhythmia e.g. chronic atrial fibrillation
    5. active pacemaker or defibrillator
12. allergy or intolerance to any of the study drugs
13. intraoperative cardiac arrhythmia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Change of intraoperative IV fentanyl consumption in the Soc+NOL guided group compared to the SoC guided group. Total consumption of fentanyl in mcg. | Intra-operative
  Change of intraoperative IV fentanyl consumption in the SoC+NOL guided group compared to the SoC guided group.
Change of frequency of intraoperative IV fentanyl administration in the Soc+NOL guided group compared to the SoC guided group. Frequency is in minutes | Intra-operative
  Change of frequency of intraoperative IV fentanyl administration in the Soc+NOL guided group compared to the SoC guided group.

SECONDARY OUTCOMES:
Change of post-operative IV hydromorphone consumption. Total consumption of hydromorphone in mcg. | PACU stay (1.5 hours)
  Change of postoperative IV hydromorphone consumption in the SoC+NOL guided group compared to the SoC guided group in the post operative care unit (PACU).
Assessment of post operative pain at rest at T0 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10 | PACU entrance
  Assessment of post operative pain at rest at T0 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at rest at T15 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10 | 15 min after PACU entrance
  Assessment of post operative pain at rest at T15 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at rest at T30 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10 | 30 min after PACU entrance
  Assessment of post operative pain at rest at T30 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at rest at T45 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10 | 45 min after PACU entrance
  Assessment of post operative pain at rest at T45 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at rest at T60 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10 | 60 min after PACU entrance
  Assessment of post operative pain at rest at T60 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at rest at T75 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10 | 75 min after PACU entrance
  Assessment of post operative pain at rest at T75 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at rest at T90 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 90 min after PACU entrance
  Assessment of post operative pain at rest at T90 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T0 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | at PACU entrance
  Assessment of post operative pain at coughing at T0 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T15 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 15 min after PACU entrance
  Assessment of post operative pain at coughing at T15 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T30 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 30 min after PACU entrance
  Assessment of post operative pain at coughing at T30 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T45 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 45 min after PACU entrance
  Assessment of post operative pain at coughing at T45 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T60 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 60 min after PACU entrance
  Assessment of post operative pain at coughing at T60 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T75 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 75 min after PACU entrance
  Assessment of post operative pain at coughing at T75 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Assessment of post operative pain at coughing at T90 minutes in PACU by using Numerical pain rating scales (NPRS) from 0 to 10. | 90 min after PACU entrance
  Assessment of post operative pain at coughing at T90 minutes in PACU by using Numerical pain rating scales (NPRS). Score is from 0 to 10.
Evaluation of intraoperative total vasoactive drugs (phenylephrine) consumption in mcg. | During anesthesia for surgery
  Evaluation of intraoperative total phenylephrine consumption (in mcg)
Evaluation of intraoperative total vasoactive drugs (ephedrine) consumption in mcg | During anesthesia for surgery
  Evaluation of intraoperative total ephedrine consumption (in mg)
Evaluation of intraoperative total vasoactive drugs (diltiazem) consumption in mg | During anesthesia for surgery
  Evaluation of intraoperative total diltiazem consumption (in mg)
Evaluation of intraoperative frequency of vasoactive drugs (phenylephrine) administration in number of events | During anesthesia for surgery
  Evaluation of intraoperative frequency of phenylephrine consumption (n)
Evaluation of intraoperative frequency of vasoactive drugs (ephedrine) administration in number of events | During anesthesia for surgery
  Evaluation of intraoperative frequency of ephedrine consumption (n)
Evaluation of intraoperative frequency of vasoactive drugs (diltiazem) administration in number of events | During anesthesia for surgery
  Evaluation of intraoperative frequency of diltiazem consumption (n)
Assessment of post operative sedation at T0 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | at PACU entrance
  Assessment of post operative sedation at T0 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Assessment of post operative sedation at T15 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | 15 min after PACU entrance
  Assessment of post operative sedation at T15 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Assessment of post operative sedation at T30 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | 30 min after PACU entrance
  Assessment of post operative sedation at T30 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Assessment of post operative sedation at T45 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | 45 min after PACU entrance
  Assessment of post operative sedation at T45 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Assessment of post operative sedation at T60 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | 60 min after PACU entrance
  Assessment of post operative sedation at T60 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Assessment of post operative sedation at T75 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | 75 min after PACU entrance
  Assessment of post operative sedation at T75 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Assessment of post operative sedation at T90 minutes in PACU by using Ramsay Sedation Score from 1 to 6 | 90 min after PACU entrance
  Assessment of post operative sedation at T90 minutes in PACU by using Ramsay Sedation Score. Score is from 1 to 6.
Number of nausea episodes in the 24 hours upon discharge from PACU | The 24 hours upon discharge from PACU
  To record the number of nausea episodes in the he 24 hours upon discharge from PACU (n)
Number of emetic episodes in the 24 hours upon discharge from PACU | The 24 hours upon discharge from PACU
  To record the number of emetic episodes (retching or vomiting) in the he 24 hours upon discharge from PACU (n)
Number of nausea AND vomiting episodes in the 24 hours upon discharge from PACU | The 24 hours upon discharge from PACU
  To record the number of nausea AND vomiting episodes in the he 24 hours upon discharge from PACU (n)
Patient self evaluation of nausea intensity | The 24 hours upon emergence
  Patient verbal rate of their worst nausea episode since emergence using a 11 points scale (0: no nausea to 10: most severe nausea)
Incidence of respiratory depression episodes | 1.5 hour since the admission to PACU
  Incidence of respiratory rate < 9 respirations per minute episodes the first 1.5 hour since the admission to PACU (n)
Incidence of requirement for naloxone reversal of opioids | 1.5 hour since the admission to PACU
  Incidence of requirement for naloxone reversal of opioids the first 1.5 hour since the admission to PACU (n)
Incidence of requirement for additional reversal of muscle relaxants | 1.5 hour since the admission to PACU
  Incidence of requirement for additional reversal of muscle relaxants the first 1.5 hour since the admission to PACU (n)
Assessment of post operative itching at T0 minutes in PACU from 0 to 10 | At PACU entrance
  Assessment of post operative itching at T0 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Assessment of post operative itching at T15 minutes in PACU from 0 to 10 | 15 min after PACU entrance
  Assessment of post operative itching at T15 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Assessment of post operative itching at T30 minutes in PACU from 0 to 10 | 30 min after PACU entrance
  Assessment of post operative itching at T30 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Assessment of post operative itching at T45 minutes in PACU from 0 to 10 | 45 min after PACU entrance
  Assessment of post operative itching at T45 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Assessment of post operative itching at T60 minutes in PACU from 0 to 10 | 60 min after PACU entrance
  Assessment of post operative itching at T60 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Assessment of post operative itching at T75 minutes in PACU from 0 to 10 | 75 min after PACU entrance
  Assessment of post operative itching at T75 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Assessment of post operative itching at T90 minutes in PACU from 0 to 10 | 90 min after PACU entrance
  Assessment of post operative itching at T90 minutes in PACU by using a 11 points scale (0: no itching, to 10: the most severe itching possible)
Post operative time to discharge from PACU in min | PACU stay (1.5 hours)
  To record the time since the admission to the discharge from PACU (min)
Time to the first postoperative pain rescue medication administration in PACU in min | PACU stay (1.5 hours)
  To record the time since the admission in the PACU to the first postoperative pain rescue medication administration in PACU (min)
Time to the first postoperative pain rescue medication administration after the PACU discharge | The 24 hours upon discharge from PACU
  To record the time since the discharge of PACU to the first postoperative pain rescue medication administration in PACU (min)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebé, MD PhD, Principal Investigator — CIUSSS Est de l'île de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal East, Quebec, Canada

REFERENCES:
- [Derived] Morisson L, Nadeau-Vallee M, Espitalier F, Laferriere-Langlois P, Idrissi M, Lahrichi N, Gelinas C, Verdonck O, Richebe P. Prediction of acute postoperative pain based on intraoperative nociception level (NOL) index values: the impact of machine learning-based analysis. J Clin Monit Comput. 2023 Feb;37(1):337-344. doi: 10.1007/s10877-022-00897-z. Epub 2022 Aug 4. PMID 35925430
- [Derived] Ghiyasinasab M, Morisson L, Laferriere-Langlois P, Geraldo-Demers MA, Gelinas C, Nadeau-Vallee M, Verdonck O, Lahrichi N, Richebe P. Identification of the intraoperative antinociceptive effect of intravenous fentanyl using the Nociception Level (NOL) index versus clinical parameters in patients undergoing gynecological laparoscopic surgery: A secondary analysis of the NOLGYN study. Anaesth Crit Care Pain Med. 2022 Aug;41(4):101102. doi: 10.1016/j.accpm.2022.101102. Epub 2022 May 25. PMID 35643392